CLINICAL TRIAL: NCT07261319
Title: Evaluating the Clinical Value of Transparent Cap-Assisted Second Examination of the Sigmoid Colon for Improving Colorectal Adenoma Detection Rates：A Single-center, Randomized Controlled Study
Brief Title: Evaluating the Clinical Value of Transparent Cap-Assisted Second Examination of the Sigmoid Colon for Improving Colorectal Adenoma Detection Rates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025K351
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Adenoma
Keywords: transparent cap; adenoma detection rate; second examination; sigmoid colon

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard second examination of the sigmoid colon (Active Comparator): Standard second examination of the sigmoid colon
  Interventions: Device: standard second examination of the sigmoid colon
- transparent cap-assisted second examination of the sigmoid colon (Experimental): transparent cap-assisted second examination of the sigmoid colon
  Interventions: Device: transparent cap-assisted second examination of the sigmoid colon

INTERVENTIONS:
Device: standard second examination of the sigmoid colon — standard second examination of the sigmoid colon
  Arms: Standard second examination of the sigmoid colon
Device: transparent cap-assisted second examination of the sigmoid colon — transparent cap-assisted second examination of the sigmoid colon
  Arms: transparent cap-assisted second examination of the sigmoid colon

SUMMARY:
A prospective, single-center, single-blind, randomized controlled study to evaluate the clinical value of transparent cap-assisted second examination of the sigmoid colon for improving colorectal adenoma detection rates

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common malignancy worldwide and the second leading cause of cancer-related mortality. In recent years, with the increasing Westernization of diet and lifestyle, the incidence and prevalence of CRC in China have risen rapidly, making CRC one of the most common gastrointestinal malignancies in the country. Its incidence and mortality now rank second and fifth, respectively, among all cancers. The disease burden of CRC in China has become substantial, and reducing its incidence and mortality is an urgent public health priority. Colonoscopy is the gold standard for CRC screening, and timely endoscopic management of precancerous lesions plays a critical role in reducing both CRC incidence and mortality.

Interval CRC refers to cancers diagnosed before the next recommended examination after a negative screening or surveillance colonoscopy. Adenoma detection rate (ADR) is an independent predictor of interval CRC risk; long-term follow-up data suggest that every 1% increase in ADR corresponds to a 5% reduction in the risk of interval CRC and a 3% reduction in mortality. However, emerging evidence indicates that interval CRC can still occur even among endoscopists with high ADRs, suggesting that some precancerous lesions may still be missed.

The main contributors to missed colorectal adenomas include: (1) operator-related factors such as fatigue, reduced attention, or limited lesion recognition; (2) image-related factors such as low-resolution visualization; and (3) inadequate mucosal exposure due to residual folds. In recent years, several studies have explored the use of "repeat intubation" to reduce missed adenomas. Multiple randomized controlled trials (RCTs) and systematic reviews have shown that a second examination can increase ADR, but most studies have focused on the right colon and often relied on chromoendoscopy or other image-enhancement modalities to improve lesion visibility. Evidence regarding second intubation specifically for the sigmoid colon remains limited, and even fewer studies have evaluated interventions based on transparent cap-assisted colonoscopy. Given that the sigmoid colon is a common site for missed polyps and adenomas, optimizing visualization in this segment may have a significant impact on overall ADR and CRC prevention.

In summary, there is still a lack of clinical evidence on whether transparent cap-assisted second intubation of the sigmoid colon can improve colorectal adenoma detection. A randomized controlled trial in the Chinese population is therefore needed to clarify its clinical value, with the potential to increase lesion detection and improve the overall quality of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* aged 45-75 years

Exclusion Criteria:

* Patients scheduled for therapeutic colonoscopy as postoperative surveillance after colorectal surgery, post-polypectomy follow-up, or treatment of histologically confirmed polyps
* Patients with highly suspected or pathologically confirmed colorectal cancer
* Patients presenting with alarm symptoms or signs (hematochezia, melena, unexplained anemia or weight loss, palpable abdominal mass, or a positive digital rectal examination)
* Pregnant or breastfeeding women
* Patients with gastrointestinal obstruction
* Patients with inflammatory bowel disease, familial adenomatous polyposis, or serrated polyposis syndrome
* Patients who have taken anticoagulants (e.g., aspirin, warfarin) within 7 days before colonoscopy or who have coagulation disorders
* Patients currently enrolled in another clinical study or who participated in any clinical trial within the past 60 days
* Insertion failure for any reason (e.g., scope cannot pass an obstruction, patient cannot tolerate the procedure) or colonoscopy not reaching the cecum
* A Boston Bowel Preparation Scale (BBPS) score < 6 at scope insertion (inadequate preparation requiring repeat bowel cleansing)
* Use of non-guideline-recommended bowel preparation agents
* Patients undergoing emergency colonoscopy
* Inadequate withdrawal time (defined as a withdrawal time <6 minutes during the first examination or <2 minutes during the second examination)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate in the rectum and sigmoid colon | 2 weeks after the procedure

SECONDARY OUTCOMES:
Increased adenoma detection rate in the rectum and sigmoid colon achieved by second examination | 2 weeks after the procedure
Adenoma miss rate in the rectum and sigmoid colon | 2 weeks after the procedure
Per-colonoscopy adenoma miss rate in the rectum and sigmoid colon | 2 weeks after the procedure
Sessile serrated lesion detection rate in rectum and sigmoid colon | 2 weeks after the procedure
Advanced adenoma detection rate in rectum and sigmoid colon | 2 weeks after the procedure
Polyp detection rate in rectum and sigmoid colon | 2 weeks after the procedure
Sessile serrated lesion detection rate | 2 weeks after the procedure
Advanced adenoma detection rate | 2 weeks after the procedure
Polyp detection rate | 2 weeks after the procedure
Perforation rate | immediately after the procedure
Clinically Significant Immediate Post-polypectomy Bleeding（CSIPB）rate | immediately after the procedure
  CSIPB was defined as any bleeding not responding to water jet irrigation or STSC and therefore requiring either coagu lation forceps or mechanical clips to achieve hemostasis
Clinically Significant Delayed Post-polypectomy Bleeding（CSDPB）rate | 2 weeks after the procedure
  CSPEB was defined as any bleeding after completion of the procedure requiring emergency room presentation, hospital isation or re-intervention (endoscopy, angiography, surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Danian Ji, Study Director — Huadong Hospital
Locations (1):
- Huadong hospital, Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: arctg4@163.com)